CLINICAL TRIAL: NCT01686321
Title: Subcutaneous Rituximab and Intravenous Bendamustine in Very Elderly Patients or Elderly Medically Non Fit Patients ("Slow Go") With Aggressive CD20-positive B-cell
Brief Title: Rituximab and Bendamustine in Very Elderly Patients or Elderly Medically Non Fit Patients With Aggressive B-cell Lymphoma
Acronym: B-R-ENDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Roche Pharma AG (Industry); Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Principal Investigator, Lorenz, Trümper, MD, Prof. Dr., University of Göttingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL-2010-1; 2010-024004-98 (EudraCT Number)
Record Dates: First submitted 2012-07-30; First posted 2012-09-18 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Aggressive Lymphoma
Keywords: elderly patients; bendamustine
MeSH Terms: interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine and subcutaneous Rituximab (Experimental): single-arm non randomized
  Interventions: Drug: Bendamustine and subcutaneous rituximab

INTERVENTIONS:
Drug: Bendamustine and subcutaneous rituximab

SUMMARY:
Bendamustine is a well tolerable and very active agent in the treatment of Non Hodgkin's lymphoma. However, in particular in aggressive B-cell lymphoma, only very few, small studies have investigated the role of bendamustine in the treatment algorithm. The aim of the current B-R-ENDA trial is to investigate efficacy and toxicity of the combination treatment of bendamustine and subcutaneous rituximab in old patients or in elderly patients with high comorbidity who do not qualify for a CHOP like treatment. The results of this study will form the basis of a larger, prospective randomized phase III trial.

DETAILED DESCRIPTION:
Bendamustine is a well tolerable and very active agent in the treatment of Non Hodgkin's lymphoma. However, in particular in aggressive B-cell lymphoma, only very few, small studies have investigated the role of bendamustine in the treatment algorithm. The aim of the current B-R-ENDA trial is to investigate efficacy and toxicity of the combination treatment of bendamustine and subcutaneous rituximab in old patients or in elderly patients with high comorbidity who do not qualify for a CHOP like treatment. The results of this study will form the basis of a larger, prospective randomized phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Histology: Diagnosis of aggressive CD20+, confirmed by an excisional biopsy of a lymph node or by a sufficiently extensive biopsy of an extranodal involvement if there is no lymph node involvement. It will be possible to treat the following entities in this study as defined by the new WHO classification of 2008: B-NHL, Follicular lymphoma grade IIIb,DLBCL, not otherwise specified (NOS),common morphologic variants: centroblastic,immunoblastic,anaplastic,rare morphologic variants.DLBCL subtypes/entities:T cell/histiocyte rich large B-cell lymphoma, primary cutaneous DLBCL, leg type, EBV-positive DLBCL of the elderly, DLBCL associated with chronic inflammation, primary mediastinal (thymic) large B-cell lymphoma, intravascular large B-cell lymphoma,ALK-positive large B-cell lymphoma, Plasmoblastic lymphoma, Primary effusion lymphoma, B-cell lymphoma, unclassifiable, with features inter¬mediate between diffuse large B-cell lymphoma and Burkitt lymphoma, B-cell lymphoma, unclassifiable, with features inter¬mediate between diffuse large B-cell lymphoma and Hodgkin lymphoma
* Stage: Any stages according to Ann Arbor Classification
* Risk group: All risk groups (IPI 1 to 5)
* Life expectancy Life expectancy of at least 6 weeks, when lymphoma is treated
* Age: Age elder than 81 or Age 61 to 80 and CIRS >6 not qualifying for CHOP-therapy
* Gender: any
* Performance status: Performance status ECOG 0 - 3. The performance status of each patient is to be assessed at the time of registration which might be after the initiation of pre-phase treatment which, as experience has shown, can result in a significant improvement of the patient´s performance status. A definition of the performance status is provided in Appendix 25.6
* Ability to give informed consent
* Written informed consent of the patient
* Contract of participation signed by the study center and sponsor

Exclusion Criteria:

* Already initiated lymphoma therapy (except for the prephase treatment until first application of rituximab)
* Serious accompanying disorder or impaired organ function (except when due to lymphoma involvement), in particular: Heart: angina pectoris CCS >2, cardiac failure NYHA >3; Lungs: the patient is to be excluded if the resultant pulmonary function test shows FEV1<50% or a diffusion capacity <50% of the reference values: Calculated creatinin clearance < 10 ml/min (Cockcroft-Gault); Liver: total bilirubin > 3 mg/dl; Uncontrollable diabetes mellitus (because of prephase treatment with prednisone!)
* Platelets <100 000/mm3, leukocytes <2500/mm3 (if not due to lymphoma)
* Known hypersensitivity to the medications to be used
* HIV-positivity
* Acute or chronic active hepatitis
* Poor patient compliance
* Simultaneous participation in other treatment studies
* Prior chemo- or radiotherapy, long-term use of corticosteroids or anti-neoplastic drugs for previous disorder
* Other concomitant tumor disease and/or tumor disease in the past 5 years (except basalioma of the skin and carcinoma in situ)
* CNS involvement of lymphoma (intracerebral, meningeal, intraspinal)
* Active serious infections not controlled by oral or intravenous antibiotics or anti-fungal
* Any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
* Non-conformity to eligibility criteria.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-07-04 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
adverse events (AE)'s | up to 30 days after last study drug administration
serious adverse events (SAE)'s | up to 30 days after last study drug administration
rate of therapy-associated deaths | up to 30 days after last study drug administration
protocol adherence | 18 weeks after start of therapy

SECONDARY OUTCOMES:
CR rate | 2 years
PR rate | 2 years
rate of primary progression | 2 years
relapse rate | 2 years
event-free survival | 2 years
overall survival | 2 years
Quality of life | 2 years
Comprehensive Geriatric Assessment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Trümper, Prof, Principal Investigator — University medicine Goettingen
Locations (1):
- Prof. Trümper, Göttingen, Germany